CLINICAL TRIAL: NCT03783182
Title: Betamethasone (Betapred®) as Premedication for Reducing Postoperative Vomiting and Pain After Tonsillectomy - a Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Betamethasone (Betapred®) as Premedication for Reducing Postoperative Vomiting and Pain After Tonsillectomy
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Eudract: 2018-001261-16
Record Dates: First submitted 2018-11-15; First posted 2018-12-20 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Tonsillectomy; Pain; PONV; Bleeding
MeSH Terms: conditions — Pain; Postoperative Nausea and Vomiting; Hemorrhage | interventions — betamethasone sodium phosphate

STUDY DESIGN:
Intervention Model Description: Double-blinded, placebo controlled and randomized study
Who Masked: Participant, Care Provider, Investigator
Masking Description: Administrator gives the study number and check the randomization list and thereafter gives the drug/placebo to a Health care personnel, who does not know if it is placebo or drug.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Betapred (Active Comparator): 16 'Betamethason Sodium Phosphate' tablets dissolved in one ml of water as part of the premedications given to the patient 30 min before the surgery
  Interventions: Drug: Betamethason Sodium Phosphate
- Placebo (Placebo Comparator): One ml of 10% glucose solution as part of the premedications given to the patient 30 min before the surgery
  Interventions: Drug: 10% glucose solution

INTERVENTIONS:
Drug: Betamethason Sodium Phosphate — Glucocorticoid
  Other Names: Betapred
  Arms: Betapred
Drug: 10% glucose solution — Glucose solution that can be used for injection, but in this case it is used perorally (one ml)
  Arms: Placebo

SUMMARY:
Betamethasone is currently given routinely in conjunction with tonsillectomy surgery at the majority of Ear, Nose & Throat clinics in Sweden. The scientific evidence regarding the effects of betamethasone in adults is limited when it comes to postoperative nausea (PONV), pain and postoperative bleeding.

DETAILED DESCRIPTION:
Steroids are used routinely aiming to reduce pain and nausea, especially in surgery with high levels of postoperative pain. The majority of international studies on tonsillectomy (TE) are performed on dexamethasone which is used in large parts of the world. Use of steroids when TE is performed on children are also more studied on than on adults. Islam et al 2011 demonstrated in a study that dexamethasone (8 mg) reduced postoperative nausea for 24 hours in a study population of both children and adults. Mc Kean et al 2006 studied the effect of 10 mg dexamethasone on nausea in adults after TE during a seven-day period. Effect was seen during the first 24 hours but not the remaining days. With regard to postoperative pain, the research results differ in terms of what effect steroids have at TE. Mc Kean et al 2006 showed significantly lower estimated pain on surgery day and day 4 to 7 after a single dose of dexamethasone peroperatively. Stewart et al 2002 has shown that, by means of preoperatively given dexamethasone (8 mg) and in decreasing dose over an 8 day period postoperative [2mgx2 for 4 days and then 2mgx1 for 4 days], the patient's estimated pain and consumption of additional pain relievers were reduced. Michele et al 1999, on the other hand, found no effect on pain over a 10 day period despite a relatively high peroperatively dose of dexamethasone (20 mg). There are, however, studies on children, suggesting that there is a dose-dependent relationship between dexamethasone and postoperative bleeding after TE in children. In a study by Czarnetzki et al 2008, 0.05, 0.15 and 0.5 mg / kg dexamethasone were used peroperatively. In this study it was seen that 0.5 mg / kg dexamethasone increased the risk of bleeding from 4% to 24%, which led to a premature termination of the study due to the bleeding risk. In 2012, a meta-analysis of the steroid effect on bleeding after tonsillectomy was conducted by Plante et al. Both studies on children and adults were included. No significant increase in the overall frequency of bleeding after tonsillectomy was seen. On the other hand, a significant increase in the number of haemorrhages that required operative action was noted. This could be interpreted as that the severity of bleedings was increased. It was recommended that systemic steroids should be used with caution until further studies have been performed. The investigators conducted a retrospective study on children with TE in Gällivare with and without betamethasone (69 patients in total) and found no evidence of increased bleeding risk, but also no effect on PONV. However, a significant effect on pain was found during the first 24 hours postoperative with the average dose of 0.15 mg / kg. When comparing different cortisone preparations, 8 mg of betamethasone corresponds to approximately 10 mg of dexamethasone. Bellis et al., 2014 performed a meta-analysis of dexamethasone and postoperative bleeding at TE in children, but considered that more studies are needed to determine the bleeding risk before any safe conclusions can be drawn. Thus, there are uncertainties with regard to the cortisone effect, both when it comes to the size of the dose and whether there really is an effect on PONV and / or postoperative pain or not. On the other hand one does not want to use high doses with risks of postoperative bleeding. Betamethasone has not been studied to the same extent as dexamethasone, and in Sweden betamethasone is preferably used preoperatively to counteract PONV and pain associated with certain operations. The results of previous studies are however not conclusive and there is no consensus of what doses that should be used. In Sweden 4 mg of betamethasone, given intravenously during the surgery, is routine at tonsillectomy surgery. However, in the literature there is very weak evidence that such a small dose have any effect. On the other hand, there are studies signaling that dexamethasone doses of 20 mg (= 16 mg betamethasone) reduced PONV, but increased postoperative hemorrhages after TE surgery.

Glucocorticoids may act via the following mechanisms: (1) anti-inflammatory effect; (2) direct central action at the solitary tract nucleus, (3) interaction with the neurotransmitter serotonin, and receptor proteins tachykinin NK1 and NK2, alpha-adrenaline, etc.; (4) maintaining the normal physiological functions of organs and systems; (5) regulation of the hypothalamic-pituitary-adrenal axis; and (6) reducing pain and the concomitant use of opioids, which in turn reduces opioid-related nausea and vomiting.

2.2. Risk/Benefit evaluation One of the main problems after tonsillectomy is PONV and especially postoperative pain that can persist up to 10-14 days after the surgery. This long period of postoperative pain leads to weakness and dehydration due to difficulties to eat and drink after the operation. Sometimes hemorrhage after TE can be fatal, but normally the bleeding can be stopped with local anaesthesia or diathermy during general anaesthesia. Normally this type of bleeding occurs in 8-10% after TE. After TE the patients normally go home the same day as the surgery. In northern Sweden the distances from the Hospital with an ear, nose and throat (ENT) emergency unit to the home of the patients could be as far as 3-400 kilometers. In this situation it is not advisory to give additional medications, which increases the risk of lethal hemorrhage.

Benefits of 8 mg betamethasone:

* Reduced PONV
* Reduced pain => Less NSAID pain killers => Less risk of hemorrhage
* Reduced pain => Increased ability to eat and drink => less risk of postoperative infection => less risk of bleeding
* Reduced pain => Shorter sick leave => Socioeconomic benefits

Risks of 8 mg betamethasone:

* Increased bleeding risk => more patients comes back to the hospital due to hemorrhage => more patients need re-surgery with diathermy of the bleeding
* Patients with gastric ulcers have an increased risk of gastric bleeding

A previous retrospective study showed a reduced pain postoperatively with 8 mg betamethasone, without any sign of increased postoperative hemorrhage. There are no studies that have showed an increased postoperative risk of hemorrhage with 10 mg of dexamethasone given to adults at TE surgery. On the other hand lower doses of dexamethasone, as for example 5 mg (= 4 mg of betamethasone), does not seem to have any clinical benefits. The aim of the present study is to evaluate if it is possible to register a beneficial effect of 8 mg betamethasone, given as a premedication orally, without increasing side effects as increased bleeding.

In conclusion, the side effects are mild and probably very infrequent, while the positive effects are visible in almost all patients with less pain and a shorter recovery period after the surgery.

3. STUDY OBJECTIVES AND ENDPOINTS 3.1. Primary objective The primary objective of this study is to verify if 8 mg of betamethasone at adolescents and adult TE operations can significantly reduce PONV.

3.2. Secondary objective(s) The secondary objective is to verify that 8 mg of betamethasone in adolescents and adult TE operations reduces postoperative pain but does not increase the postoperative bleeding risks.

4. STUDY DESIGN AND PROCEDURES 4.1. Overall study design and flow chart

The study is a double-blind, placebo-controlled, randomized study in 100 volunteered patients over 12 years of age selected for elective tonsillectomy at the ENT clinic in Norrbotten. Patients fulfilling all of the inclusion and none of the exclusion criterias will be included. Enrollment will be continued until the required sample size is achieved (100 subjects). Once informed consent is obtained, screening data will be collected to determine each subject´s eligibility for study participation. The total expected duration of the subject participation is maximum 95 days, from screening visit to end of follow-up. The active participation is 5 days (surgery at visit 2 and phone calls, 1 and 5 days after day of surgery). The study pharmaceutical (betamethasone) is a well-known substance and has been used in humans for many years for the same indications as in the present study. Thus it will be regarded as a phase IV study.

ELIGIBILITY:
Inclusion Criteria:

Signed informed consent Age over 12 years Planned for elective bilateral tonsillectomy

Exclusion Criteria:

* • Insulin dependent diabetes mellitus

  * NSAID or corticosteroid intolerance
  * Pregnancy
  * Gastric ulcer
  * Immunodeficiency
  * Treatment for chronic pain
  * Psychiatric disorders

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-09-10 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Postoperative nausea and vomiting | 0-5 days postop
  Nausea/Vomiting postoperatively, numeric Visual Analogue Scale graded from 0 to 10, where 10 is the worst grade of nausea

SECONDARY OUTCOMES:
Postoperative pain | 0-5 days postop
  Postoperative pain, numeric Visual Analogue Scale, graded from 0 to 10, where grade 10 is the worse pain

OTHER OUTCOMES:
Postoperative bleeding | 0-30 days postop
  Postoperative bleeding, visits to Health care. Medical records of the patients are used retrospectively in order to detect any postoperative bleeding that has caused a Contact with the Health care. Such events are divided in a) no of events not demanding new surgery and b) no of events demanding hemostasis by new surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Krister Tano, MD, PhD, Principal Investigator — Umeå University
Locations (1):
- Sunderby sjukhus, Luleå, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Islam MR, Haq MF, Islam MA, Meftahuzzaman SM, Sarkar SC, Rashid H, Rashid HU. Preoperative use of granisetron plus dexamethasone and granisetron alone in prevention of post operative nausea and vomiting in tonsillectomy. Mymensingh Med J. 2011 Jul;20(3):386-90. PMID 21804499
- [Background] McKean S, Kochilas X, Kelleher R, Dockery M. Use of intravenous steroids at induction of anaesthesia for adult tonsillectomy to reduce post-operative nausea and vomiting and pain: a double-blind randomized controlled trial. Clin Otolaryngol. 2006 Feb;31(1):36-40. doi: 10.1111/j.1749-4486.2006.01141.x. PMID 16441800
- [Background] Stewart R, Bill R, Ullah R, McConaghy P, Hall SJ. Dexamethasone reduces pain after tonsillectomy in adults. Clin Otolaryngol Allied Sci. 2002 Oct;27(5):321-6. doi: 10.1046/j.1365-2273.2002.00588.x. PMID 12383289
- [Background] Carr MM, Williams JG, Carmichael L, Nasser JG. Effect of steroids on posttonsillectomy pain in adults. Arch Otolaryngol Head Neck Surg. 1999 Dec;125(12):1361-4. doi: 10.1001/archotol.125.12.1361. PMID 10604415
- [Background] Czarnetzki C, Elia N, Lysakowski C, Dumont L, Landis BN, Giger R, Dulguerov P, Desmeules J, Tramer MR. Dexamethasone and risk of nausea and vomiting and postoperative bleeding after tonsillectomy in children: a randomized trial. JAMA. 2008 Dec 10;300(22):2621-30. doi: 10.1001/jama.2008.794. PMID 19066382
- [Background] Plante J, Turgeon AF, Zarychanski R, Lauzier F, Vigneault L, Moore L, Boutin A, Fergusson DA. Effect of systemic steroids on post-tonsillectomy bleeding and reinterventions: systematic review and meta-analysis of randomised controlled trials. BMJ. 2012 Aug 28;345:e5389. doi: 10.1136/bmj.e5389. PMID 22930703
- [Background] Johansson U, Sundgren C, Tano K, van den Berg J. The effect of Perioperative Bethamethasone on Post-operative Nausea, Vomiting and Pain in Children undergoing Tonsillar Surgery. British Journal of Anaesthetic&Recovery Nursing. 2011;11:24-29.
- [Background] Bellis JR, Pirmohamed M, Nunn AJ, Loke YK, De S, Golder S, Kirkham JJ. Dexamethasone and haemorrhage risk in paediatric tonsillectomy: a systematic review and meta-analysis. Br J Anaesth. 2014 Jul;113(1):23-42. doi: 10.1093/bja/aeu152. PMID 24942713
- [Background] Chu CC, Hsing CH, Shieh JP, Chien CC, Ho CM, Wang JJ. The cellular mechanisms of the antiemetic action of dexamethasone and related glucocorticoids against vomiting. Eur J Pharmacol. 2014 Jan 5;722:48-54. doi: 10.1016/j.ejphar.2013.10.008. Epub 2013 Nov 1. PMID 24184695